CLINICAL TRIAL: NCT00005944
Title: Study of Second Look Surgery With or Without Chemotherapy Intraperitoneally, in the Event of Risk of Intraperitoneal Recurrence
Brief Title: Second-look Surgery With or Without Intraperitoneal Chemotherapy in Treating Patients With Recurrent Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insuffisient recruitment
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067833; FRE-FNCLCC-97018; EU-20010
Record Dates: First submitted 2000-07-05; First posted 2004-03-24 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer; Metastatic Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases; primary peritoneal cavity cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Drug Therapy; Fluorouracil; Leucovorin; Mitomycin; Laparoscopy

INTERVENTIONS:
Drug: chemotherapy
Drug: fluorouracil
Drug: leucovorin calcium
Drug: mitomycin C
Procedure: conventional surgery
Procedure: laparoscopic surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs in different ways may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of second-look surgery with or without intraperitoneal infusions of mitomycin and fluorouracil in treating patients who have colorectal cancer that is recurrent to the peritoneum.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the effect of second look surgery with or without intraperitoneal mitomycin and fluorouracil on the 3 year survival rate of patients with colorectal cancer who are at high risk for peritoneal cavity cancer. II. Compare the quality of life of patients treated with these regimens. III. Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, risk group, presence of symptoms (yes vs no), and isolated disease (yes vs no). After primary surgery, all patients receive 6 months of chemotherapy consisting of leucovorin calcium IV followed by fluorouracil IV over 10 minutes on days 1-5 every 4 weeks. Patients then undergo second look surgery or laparoscopy at 8-12 months. Second look surgery or laparoscopy may be performed earlier if markers increase progressively for unknown reasons or symptoms of peritoneal cancer occur. Patients with recurrent disease that can be resected are randomized to one of two treatment arms. Patients with no residual disease or with unresectable disease are followed for survival. Arm I: Patients undergo complete resection of all detectable lesions followed immediately by intraperitoneal (IP) mitomycin on day 0 and fluorouracil IP on days 1-4. Patients also receive systemic chemotherapy consisting of leucovorin calcium IV over 2 hours and fluorouracil IV bolus, followed by fluorouracil IV over 22 hours on days 1 and 2. Systemic chemotherapy repeats every 2 weeks for 6 months. Arm II: Patients undergo complete or partial resection and then receive systemic chemotherapy as in arm I. Quality of life is assessed at baseline and then every 4 months for 3 years. All patients (including nonrandomized patients) are followed every 4 months for 3 years.

PROJECTED ACCRUAL: A total of 152 patients (76 randomized) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Primary diagnosis of adenocarcinoma of the colon or rectum and meeting one of the following risk criteria during the primary surgery: Perforated bowel (spontaneous or not) Occlusion Peritoneal deposits Invasion of serosa of more than 4 cm diameter Concurrent ovarian metastases Randomization eligibility: Presence of proven recurrent peritoneal disease (only one micronodule of 1 mm sufficient) at second look laparotomy Total resection of macroscopic lesions possible (local recurrence, lymph node or hepatic metastases)

PATIENT CHARACTERISTICS: Age: 70 and under Performance status: Not specified Life expectancy: Not specified Hematopoietic: WBC at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 1.4 mg/dL Cardiovascular: No cardiac condition that would increase surgical risk Pulmonary: No pulmonary condition that would increase surgical risk Other: No other condition that would increase surgical risk No other malignancy within the past 5 years except basal cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: No concurrent anticancer radiotherapy Surgery: See Disease Characteristics

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07-01 (Actual); Primary Completion 2000-10-24 (Actual); Study Completion 2003-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Elias, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (18):
- CHU Sart-Tilman, Liège, Belgium
- France (17):
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier Regional de Lille, Lille
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHR Hotel Dieu, Nantes
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Hopital L'Archet - 2, Nice
  - C.H.R. de Nimes - Hopital Caremeau, Nîmes
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Centre Hospitalier Universitaire, Reims
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif